CLINICAL TRIAL: NCT03001466
Title: A Randomized Controlled Trial Comparing Urea Loaded Nanoparticles to Placebo: a New Concept for Cataract Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Mohamed Saad Eldien, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NCCM
Record Dates: First submitted 2016-10-01; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Drug Action Increased
Keywords: Cataract; Urea-loaded NPs; TEM examination
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- urea-loaded nanoparticles eye drops (Experimental): This arm include 40 cases (67 eyes) received urea-loaded nanoparticles eye drops (one drop five times a day for 8 weeks)
  Interventions: Drug: urea-loaded nanoparticles eye drops
- Balance Salt Solution eye drops (Placebo Comparator): This arm include 11 cases (22 eyes) recieved Balance Salt Solution eye drops (one drop five times a day for 8 weeks)
  Interventions: Drug: Balance Salt Solution eye drops

INTERVENTIONS:
Drug: urea-loaded nanoparticles eye drops — one drop five times a day for 8 weeks
  Other Names: pluronic®F-127 (PF)
  Arms: urea-loaded nanoparticles eye drops
Drug: Balance Salt Solution eye drops — one drop five times a day for 8 weeks
  Other Names: Balance Salt Solution
  Arms: Balance Salt Solution eye drops

SUMMARY:
Cataract is the leading cause of vision loss and blindness in the world,surgery is the only available option to correct the problem and the major reasons for low cataract surgical rates include low demand because of fear of surgery, high cost of surgery and poor visual results but new research raises the hope that someday, cataracts could be cured with simple eye drops. This is the first report for preparing urea-loaded NPs eye drops for cataract therapy. Enhancement of the urea efficacy is accomplished by using polymeric NPs based on the amphiphilic block copolymer Pluronic®F-127 (PF) which is a hydrophilic nontoxic copolymer widely used as a pharmaceutical excipient for its stabilizing properties and capability to increase the solubility.

DETAILED DESCRIPTION:
51 patients with cataract were included in this study that started at December 2014 to April 2016. All cases collected from out patients' clinic of Assiut University Hospital These patients were randomized into two groups. Group I(control) included 11 cases (22 eyes) used Balance Salt Solution (BSS) eye drops. Group II include 40 cases (67 eyes) were treated by the prepared eye drops of urea NPs solution.

Preparation of urea-loaded nanoparticles

First the investigators will test the safety of urea as eye drops by injecting urea in concentration of 96 ml/mol in the anterior chamber of 6 rabbit eyes and the other eye of each rabbit will be used as control. After 14 days enucleation of both eyes, then will prepare extracted eye tissue for examination by light and electron microscopes.

Urea solution will be then prepared for eye drops purpose by enhancing its efficacy using the polymeric NPs based on the amphiphilic block copolymer Pluronic®F-127 (PF) which is an A-B-A-type triblock copolymer consisting of polyoxyethylene (PEO) units (A) and polyoxypropylene (PPO) units (B) with a thermoreversible gelation property that has a hydrophilic nontoxic property widely used as a pharmaceutical excipient for its stabilizing properties and capability to increase the solubility.

The eye drop will be prepared by an ionic gelation method using the tripeptide antioxidant glutathione (GSH) with the pluronic®F-127 (PF) as carriers to urea delivery for the target of cataract therapy. Pluronic® F127 (PF127), which can be self-assembled into micelles upon increasing concentration or raising temperatures, is used to decorate the water-soluble urea via a chemical reaction. Next, the GSH is incorporated into the hydrophobic poly (propylene oxide) compartment of PF127 using electrostatic interactions between the positively charged GSH and the negatively charged PF. The prepared NPs were then characterized using transmission electron microscopy (TEM). The average size of urea-loaded PF 127/GSH NPs was 140 nm.

ELIGIBILITY:
Inclusion Criteria:

* All cases were immature cataract at different stages.

Exclusion Criteria:

* No complicated cataract included in this study either due to local or systemic diseases.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
the difference in the score of visual acuity. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hassan L Fahmy, Prof, Principal Investigator — Assiut university-Faculty of medicine

IPD SHARING:
Plan to Share IPD: No